CLINICAL TRIAL: NCT06422598
Title: Prevalence and Management Practice of Diabetic Kidney Disease at BADAS Affiliated Healthcare Centres in Bangladesh - An Exploratory Cross-Sectional Study
Brief Title: Prevalence and Management Practice of Diabetic Kidney Disease at BADAS Affiliated Healthcare Centres in Bangladesh
Acronym: BADAS
Status: Recruiting | Type: Observational
Sponsor: Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders (Other)
Collaborators: Ibrahim Medical College (Unknown)
Responsible Party: Principal Investigator, Wasim Md Mohosin Ul Haque, Professor, Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders
Other Study IDs: BADAS-ERC/EC/24/23; BADAS-ERC/EC/24/23 (Other: The Diabetic Association of Bangladesh (BADAS))
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Kidney Disease
Keywords: diabetes; Diabetic kidney disease; Prevalence; management
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Diabetes is a growing public health concern in Bangladesh, with millions affected. Diabetic Kidney Disease (DKD) is a severe complication of diabetes, affecting approximately 21.3% of the diabetic population. To address this issue, a comprehensive assessment of DKD within the Bangladesh Diabetic Association's (BADAS) affiliated healthcare centres is necessary.

Objective: The study's general objective is to determine the prevalence of DKD and evaluate its management at BADAS-affiliated healthcare centers. Specific objectives include assessing risk factors, screening practices, disease staging, management approaches, patient education, and providing evidence-based recommendations.

Methodology:

* Study Design: Cross-sectional
* Study Population: All diabetic patients at BADAS-affiliated centers
* Exclusion Criteria: Patients unwilling to participate or with kidney disease from other causes and with acute illness
* Sample Size: "Forty patients will be selected from each center, resulting in a total sample size of 320 patients across eight centers, with one center randomly selected from each of the eight divisions in Bangladesh."
* Data Collection: Demographics, comorbidities, kidney function, blood pressure, HbA1c levels, medication records, treatment guideline adherence
* Data Analysis: prevalence of diabetic kidney disease, factors affecting management, and potential barriers
* Ethical Considerations: Ensure patient data privacy, obtain approvals, and informed consent Implications: The study aims to provide insights into the current state of magnitude (prevalence) of DKD, its management, highlighting areas for improvement in patient care, guideline adherence, and ultimately enhancing the well-being of diabetic patients in Bangladesh.

DETAILED DESCRIPTION:
Background: Diabetes mellitus represents a significant public health challenge globally, and Bangladesh is no exception to this growing epidemic. According to the International Diabetes Federation (IDF), about 13.1 million people in Bangladesh have diabetes, and this number is expected to increase to 22.3 million by 2045(Sun et al., 2022). One of the most serious complications of diabetes is Diabetic Kidney Disease (DKD), which can lead to chronic kidney disease and end-stage renal disease (ESRD). DKD not only imposes a heavy burden on the healthcare system but also affects the economic and social well-being of the patients and their families. The prevalence of kidney disease among the diabetic population of Bangladesh is estimated to be around 21.3%. This number is based on a single center study conducted at the Bangladesh Institute of Health Sciences (BIHS) hospital in Dhaka, Bangladesh(Islam et al., 2021). This high prevalence highlights the need for a comprehensive evaluation of DKD within the centers affiliated with the Bangladesh diabetic association (BADAS), which is the largest non-governmental organization providing diabetes care and research in the country.

The Bangladesh Diabetic Association (BADAS), with its extensive network of diabetes care centers and healthcare professionals, has long been at the forefront of addressing diabetes-related health concerns in the country. As a nation-wide institution dedicated to diabetes care, BADAS plays a pivotal role in delivering healthcare services and shaping the well-being of diabetic patients in Bangladesh.

A comprehensive understanding of DKD prevalence and management status within BADAS centers is essential to enhance the quality of care for diabetic patients. Identifying areas for improvement is the first step towards effecting positive change.

Our ultimate plan is to implement a nationwide DKD prevention program through affiliated diabetic centers. To achieve this, a comprehensive assessment of the current situation is an imperative foundation for program design, planning, and execution.

The study will provide a rich dataset upon which evidence-based recommendations for preventing and managing DKD within BADAS-affiliated centers can be developed. These recommendations are essential for improving patient outcomes and ensuring the success of the future prevention program.

In conclusion, the proposed study is a crucial undertaking aimed at addressing the pressing issue of DKD within the context of BADAS-affiliated healthcare centers. It serves as the first step towards the larger goal of implementing a nationwide DKD prevention program, with the potential to positively impact the health and well-being of diabetic patients across Bangladesh.

Objective:

General Objective:

To determine the prevalence of diabetic kidney disease and assess the management status of diabetic kidney disease in patients attending affiliated healthcare centers of the Bangladesh Diabetic Associations.

Specific Objectives:

Determine the Prevalence of Diabetic Kidney Disease: Calculate the prevalence of DKD among diabetic patients visiting BADAS-affiliated healthcare centers using clinical and laboratory assessments.

Assess Risk Factors for DKD: Identify and analyze demographic and clinical factors associated with the development of DKD in the study population.

Evaluate Screening Practices: Evaluate the extent to which BADAS-affiliated healthcare centers conduct regular screening of registered diabetic patients for DKD and assess the effectiveness of current screening protocols.

Characterize Disease Staging: Determine the stages of DKD among patients diagnosed with the condition and assess the proportion of patients with various stages of renal impairment.

Analyze Management Approaches: Investigate the treatment modalities, including pharmacological interventions, lifestyle modifications, and patient education, used to manage DKD in the healthcare centers.

Assess Healthcare Professional Awareness: Evaluate the awareness and knowledge of healthcare professionals working in BADAS-affiliated centres regarding DKD prevention, diagnosis, and management.

Assess the infrastructural support of BADAS-affiliated centres regarding DKD prevention, diagnosis, and management.

Examine Patient Education and Engagement: Assess the level of patient education and engagement in DKD management programs, including lifestyle modification guidance and adherence to treatment plans.

Provide Recommendations: Based on the study findings, generate evidence-based recommendations for improving the prevention, early detection, and management of DKD in BADAS-affiliated healthcare centers to enhance the quality of care for diabetic patients.

Material and Methodology:

Study Design:

Cross-sectional study design.

Study Population:

All registered diabetic patients receiving care at affiliated healthcare centres of Bangladesh Diabetic Associations.

Exclusion criteria:

Unwilling to participate in the study. Presence of AKI or acute illness Presence of Known kidney disease due to other cause.

Sampling method: Multi-stage sampling.

Sample size calculation:

The formula to calculate the sample size:

Where:

n = required sample size Z = Z-score corresponding to the desired confidence level (e.g., 1.96 for a 95% confidence level) p = expected prevalence (in decimal form) E = margin of error (in decimal form) Expected prevalence of DKD to be 21.3% (0.213 in decimal form) Confidence level 95% Margin of error of 5% (0.05 in decimal form)

Using these values, the sample size calculation would look like this:

= 292 However, we will select forty patients from each centre, resulting in a total sample size of 320 patients across eight centres, with one centre will be randomly selected from each of the eight divisions in Bangladesh.

Data Collection:

Gather patient data, including demographics, comorbidities, kidney function (eGFR, UACR), blood pressure measurements, and HbA1c levels.

Review medication records to determine the use of anti-proteinuric medications (e.g., ACE inhibitors, angiotensin receptor blockers, SGLT2i, nonsteroidal mineralocorticoids receptor antagonists and GLP analogues).

Assess adherence to recommended treatment guidelines for diabetic kidney disease management.

Collect data on healthcare professionals' awareness and knowledge of DKD prevention, diagnosis, and management.

Gather data on the infrastructure available in BADAS-affiliated centres for DKD prevention, diagnosis, and management.

Screening for the presence of DKD

The diagnostic criteria for diabetic kidney disease (DKD)(McGrath and Edi, 2019, ElSayed et al., 2022):

DKD is usually a clinical diagnosis in a patient with long-standing diabetes (>10 years) with albuminuria and/or reduced eGFR in the absence of signs or symptoms of other primary causes of kidney damage.

Albuminuria: Increased urinary albumin excretion is defined as ≥30 mg/g. (2 out of 3 in 3 to 6 months).

Reduced estimated Glomerular Filtration Rate (eGFR): <60ml/minute/1.73m2. for more than 3 months Duration of Diabetes: DKD is typically associated with a long duration of diabetes (>10 years' duration of type 1 diabetes; may be present at diagnosis in type 2 diabetes).

Presence of Retinopathy: DKD is typically associated with retinopathy however the absence of retinopathy does not exclude DKD in type 2 diabetes.

Data Analysis:

Evaluate the proportion of patients achieving target blood pressure control (e.g., <130/80 mm Hg), glycaemic control (e.g., HbA1c <7%), and receiving appropriate anti-proteinuric medications.

Examine factors associated with successful management, including age, gender, duration of diabetes, and comorbidities.

Identify potential barriers to achieving optimal management.

Ethical Considerations:

Ensure patient data privacy and confidentiality. Obtain necessary approvals and informed consent for data access and analysis.

Implications:

Provide insights into the current magnitude and state of diabetic kidney disease management, specifically focusing on blood pressure and glycaemic control and the utilization of anti-proteinuric medications among diabetic patients.

Highlight areas for improvement in patient care and guideline adherence to enhance diabetic kidney disease management.

ELIGIBILITY:
Inclusion Criteria:

• All registered diabetic patients receiving care at affiliated healthcare centres of Bangladesh Diabetic Associations.

Exclusion Criteria:

* Unwilling to participate in the study.
* Presence of AKI or acute illness
* Presence of Known kidney disease due to other cause.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will select forty patients from each centre, resulting in a total sample size of 320 patients across eight centres, with one centre will be randomly selected from each of the eight divisions in Bangladesh
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2024-05-11 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of diabetic kidney disease | Day 1
  Calculate the prevalence of DKD among diabetic patients visiting BADAS-affiliated healthcare centers using clinical and laboratory assessments.

SECONDARY OUTCOMES:
Risk Factors for DKD | Day 1
  Identify and analyze demographic and clinical factors associated with the development of DKD in the study population.
Screening Practices | Day 1
  Evaluate the extent to which BADAS-affiliated healthcare centers conduct regular screening of registered diabetic patients for DKD and assess the effectiveness of current screening protocols.
Management Approaches | Day 1
  Investigate the treatment modalities, including pharmacological interventions, lifestyle modifications, and patient education, used to manage DKD in the healthcare centers.

CONTACTS AND LOCATIONS:
Overall Officials: Wasim MM Haque, MBBS, FCPS, Principal Investigator — Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders
Locations (8):
- Bangladesh (8):
  - Chapainawabganj Diabetes Center, Chapainawabganj
  - Cox's Bazar Diabetic Hospital, Cox’s Bāzār
  - Meherpur diabetes hospital, Meherpur
  - Narayanganj Diabetic Hospital, Nārāyanganj
  - Diabetic Hospital Panchagarh, Panchagarh
  - Pirojpur Diabetic Samiti, Pirojpur
  - Rajbari Diabetes Center, Rājbāri
  - Sherpur Diabetic Hospital, Sherpur

REFERENCES:
- [Result] ElSayed NA, Aleppo G, Aroda VR, Bannuru RR, Brown FM, Bruemmer D, Collins BS, Hilliard ME, Isaacs D, Johnson EL, Kahan S, Khunti K, Leon J, Lyons SK, Perry ML, Prahalad P, Pratley RE, Jeffrie Seley J, Stanton RC, Gabbay RA, on behalf of the American Diabetes Association. 15. Management of Diabetes in Pregnancy: Standards of Care in Diabetes-2023. Diabetes Care. 2023 Jan 1;46(Suppl 1):S254-S266. doi: 10.2337/dc23-S015. PMID 36507645
- [Result] Islam SMS, Salehin M, Zaman SB, Tansi T, Gupta RD, Barua L, Banik PC, Uddin R. Factors Associated with Chronic Kidney Disease in Patients with Type 2 Diabetes in Bangladesh. Int J Environ Res Public Health. 2021 Nov 23;18(23):12277. doi: 10.3390/ijerph182312277. PMID 34886001
- [Result] McGrath K, Edi R. Diabetic Kidney Disease: Diagnosis, Treatment, and Prevention. Am Fam Physician. 2019 Jun 15;99(12):751-759. PMID 31194487
- [Result] Sun H, Saeedi P, Karuranga S, Pinkepank M, Ogurtsova K, Duncan BB, Stein C, Basit A, Chan JCN, Mbanya JC, Pavkov ME, Ramachandaran A, Wild SH, James S, Herman WH, Zhang P, Bommer C, Kuo S, Boyko EJ, Magliano DJ. IDF Diabetes Atlas: Global, regional and country-level diabetes prevalence estimates for 2021 and projections for 2045. Diabetes Res Clin Pract. 2022 Jan;183:109119. doi: 10.1016/j.diabres.2021.109119. Epub 2021 Dec 6. PMID 34879977